CLINICAL TRIAL: NCT03520387
Title: Combined Treatments to Optimize Functional Recovery in Veterans With Chronic Low Back Pain
Brief Title: Selecting Effective Combinations of Treatment for Low Back Pain
Acronym: SELECT LBP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: F2891-P
Record Dates: First submitted 2018-04-27; First posted 2018-05-09 (Actual); Results first posted 2021-09-05 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-08

CONDITIONS: Low Back Pain
Keywords: Randomized controlled trial; Chronic pain
MeSH Terms: conditions — Low Back Pain; Chronic Pain | interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: The proposed research assesses the feasibility of using a 2 x 2 factorial randomized controlled trial (RCT) design to examine the individual and combined effects of 1) lumbar medial branch nerve radiofrequency ablation (LRFA) (vs. simulated LRFA control), and 2) a novel video telehealth tablet- and personal computer (PC)-based Activity Tracker-Informed Video-Enabled Cognitive Behavioral Therapy program ("AcTIVE-CBT") (vs. a telephone-based self-directed CBT and education control). This pilot RCT will involve 30 Veterans with chronic low back pain (CLBP) who will be followed to evaluate functional recovery for 3 months.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Some investigators are not masked, for safety monitoring purposes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Lumbar medial branch nerve radiofrequency ablation (LRFA) (Experimental): Radiofrequency ablation of the dorsal rami of the lumbar spinal nerves
  Interventions: Procedure: Lumbar medial branch nerve radiofrequency ablation (LRFA)
- Simulated lumbar radiofrequency ablation (simulated LRFA) (Active Comparator): Simulated radiofrequency ablation of the dorsal rami of the lumbar spinal nerves(simulated LRFA), with targeted steroid injections
  Interventions: Procedure: Simulated LRFA with targeted steroid injections
- AcTIVE-CBT (Experimental): Activity-Tracker Informed Video-enabled Cognitive Behavioral Therapy (AcTIVE-CBT)
  Interventions: Behavioral: AcTIVE-CBT
- TBSCE (Active Comparator): Telephone-based self-directed CBT and education (TBSCE)
  Interventions: Behavioral: TBSCE

INTERVENTIONS:
Procedure: Lumbar medial branch nerve radiofrequency ablation (LRFA) — Radiofrequency ablation of the dorsal rami of the lumbar spinal nerves, using electrode placement parallel to the medial branches, 18G electrodes or larger, and 2 lesions per nerve.
  Arms: Lumbar medial branch nerve radiofrequency ablation (LRFA)
Procedure: Simulated LRFA with targeted steroid injections — Performed in an identical fashion to the experimental arm (LRFA), except for medial branch lesioning, which will not be done in simulated LRFA, and 2) the simulated LRFA control group will receive an injection of triamcinolone acetonide at each site where a radiofrequency lesion would normally be applied.
  Other Names: Simulated radiofrequency ablation of the dorsal rami of the lumbar spinal nerves(simulated LRFA), with targeted steroid injections to the medial branch nerves.
  Arms: Simulated lumbar radiofrequency ablation (simulated LRFA)
Behavioral: AcTIVE-CBT — AcTIVE-CBT involves a standardized CBT protocol for pain, delivered via a video telehealth interface. AcTIVE-CBT also incorporates use of an activity tracker to provide objective feedback on activity levels, which can inform participants' and providers' impressions of goals and progress.
  Other Names: Activity-Tracker Informed Video-enabled Cognitive Behavioral Therapy (AcTIVE-CBT).
  Arms: AcTIVE-CBT
Behavioral: TBSCE — TBSCE control is a focused program of CBT involving an initial 60-minute telephone education session by a psychologist; the provision of printed educational materials on chronic pain self-management, and a workbook for CBT self-management; and structured, written plans for weekly practice, reading and homework using the workbook.
  Other Names: Telephone-based supportive contact and education (TBSCE)
  Arms: TBSCE

SUMMARY:
Back pain is the #1 contributor to disability in the United States (US), and second only to hearing problems as a reason for new Veteran disability compensation. The societal burden of back pain is driven mainly by chronic low back pain (CLBP), defined as low back pain persisting for 3 months. Since most individual treatments for CLBP have only small effects on functional recovery, combining CLBP treatments has recently been recommended as a priority area for research. However, few prior studies of CLBP have been properly designed to evaluate the effects of treatment combinations. Large effects on functional recovery from CLBP may require combining interventions that each target different points on a theoretical pathway to functional recovery. Procedural treatments for CLBP aim primarily to address early stages in the pathway to functional recovery, such as problems with the lumbar spinal structures or low back pain itself. In contrast, behavioral interventions for CLBP generally have effects not only on pain itself, but also work by mitigating the degree to which the sensation of low back pain impacts function, well-being, and quality of life. These represent later stages in the pathway to functional recovery from CLBP. Combining procedural and behavioral treatments may have great potential for achieving large magnitude treatment effects for CLBP in Veterans.

The proposed research assesses the feasibility of using a 2 x 2 factorial randomized controlled trial (RCT) design to examine the individual and combined effects of 1) lumbar medial branch nerve radiofrequency ablation (LRFA), a commonly used procedural intervention to target low back pain severity, and 2) a novel video telehealth tablet- and personal computer (PC)-based Activity Tracker-Informed Video-Enabled Cognitive Behavioral Therapy program ("AcTIVE-CBT"), a behavioral intervention designed primarily to target functional limitations both secondary to, and independent of, improvements in pain. The LRFA treatment to be used in the proposed study addresses the major patient selection, procedural/technical, methodologic and reporting limitations of prior studies. AcTIVE-CBT addresses problems with Veteran access and compliance associated with conventional cognitive behavioral therapy (CBT) delivered in clinic, and uses currently available activity tracking technology to better promote activity and behavior change as compared to conventional CBT. This pilot RCT involves recruitment of up to 30 Veterans with CLBP who will be followed to evaluate functional recovery for up to 3 months, to reach a goal of 20 Veterans completing the 3-month primary outcome. The primary outcome is participant-reported back-related functional limitations (mobility and ADLs) at 3 months, as measured by the validated Roland-Morris Disability Questionnaire. Secondary outcomes include activity tracker-assessed step counts, back pain intensity, reduction in opioid use, and quality of life. Although the proposed pilot study is unlikely to definitively address whether these treatments alone or in combination have significant effects on functional recovery, it will inform a future large-scale multicenter RCT to determine the efficacy of LRFA, AcTIVE-CBT, or combined LRFA + AcTIVE-CBT, for Veterans with CLBP.

DETAILED DESCRIPTION:
The proposed research assesses the feasibility of using an innovative application of the 2 x 2 factorial randomized controlled trial (RCT) design to examine the individual and combined effects of 1) lumbar medial branch nerve radiofrequency ablation (LRFA), a commonly used procedural intervention to target low back pain severity, and 2) a novel video telehealth tablet- and personal computer (PC)-based Activity Tracker-Informed Video-Enabled Cognitive Behavioral Therapy program ("AcTIVE-CBT"), a behavioral intervention designed primarily to target functional limitations both secondary to, and independent of, improvements in pain. The LRFA treatment to be used in the proposed study addresses the major patient selection, procedural/technical, methodologic and reporting limitations of prior studies. AcTIVE-CBT addresses problems with Veteran access and compliance associated with conventional cognitive behavioral therapy (CBT) delivered in clinic, and uses currently available activity tracking technology to better promote activity and behavior change as compared to conventional CBT. This pilot RCT involves recruitment of up to 30 Veterans with CLBP who will be followed to evaluate functional recovery for up to 3 months, to reach a goal of 20 Veterans completing the 3-month primary outcome. The primary outcome is participant-reported back-related functional limitations (mobility and ADLs) at 3 months, as measured by the validated Roland-Morris Disability Questionnaire. Secondary outcomes include activity tracker-assessed step counts, back pain intensity, reduction in opioid use, and quality of life. The investigators hypothesize that 1) each individual treatment will result in improvements in back-related functional limitations and secondary outcomes compared to control, and 2) combined treatment will produce greater treatment effects than each of the individual treatments alone. Although the proposed pilot study is unlikely to definitively address whether these treatments alone or in combination have significant effects on functional recovery, it will inform a future large-scale multicenter RCT to determine the efficacy of LRFA, AcTIVE-CBT, or combined LRFA + AcTIVE-CBT, for Veterans with CLBP.

ELIGIBILITY:
Inclusion Criteria:

* Adult Veteran seeking care in the VA Puget Sound Health Care System
* Chronic low back pain of duration at least 3 months
* Low back pain intensity numerical rating scale (NRS) 4 (must be 4 or higher)
* Has failed 1st line rehabilitative treatments, including physical therapy, yoga, tai chi, chiropractic or osteopathic manipulation, and/or massage.
* Must be able to provide informed consent and complete the assessment instruments accurately
* Must have access to a computer, tablet, or smartphone with internet access at home or at work
* 'Positive responses' to 2 separate sets of lumbar medial branch blocks (MBBs: low volume anesthetic blocks of the medial branches of the dorsal rami using 0.5cc or less of lidocaine or bupivacaine), including at least 50% pain improvement of typical low back pain, with onset of typical lumbar back pain relief within 30 mins and relief lasting at least 30 mins after the onset of initial pain relief
* Considered a candidate for unilateral or bilateral LRFA at 2-4 spinal levels (between L1 and S1)

Exclusion Criteria:

* Clinical suspicion that the current low back pain symptoms have a significant and sustained component that is attributed to specific lumbar spine-related syndromes including lumbosacral radicular syndrome (radiculopathy), symptomatic lumbar spinal stenosis (neurogenic claudication), with confirmatory imaging findings, spinal instability requiring surgery, or 'red flag' conditions (infection/ malignancy/ fracture)
* Pregnant females, prisoners, or the cognitively impaired
* Prior lumbar RFA
* Prior lumbar spine surgery involving the levels where LRFA is to be performed, within the past 2 years
* Lumbar fusion or instrumentation involving the levels where LRFA is to be performed
* Prior CBT for chronic pain
* Primary psychotic or major thought disorder (lifetime), any active suicidal/homicidal ideation (past 6 months), unstable or severe psychiatric/behavioral conditions (e.g. delirium, mania, psychosis)
* Hospitalization for psychiatric reasons involving psychosis other than suicidal ideation, homicidal ideation, and/or PTSD, in the past 5 years
* Cognitive limitations that would prevent participation
* Severe medical comorbidities posing major functional limitations in ambulation and function or medical prognosis, including vascular, pulmonary or coronary artery disease, metastatic cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2018-11-15 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pradeep Suri, MD, Principal Investigator — VA Puget Sound Health Care System Seattle Division, Seattle, WA
Locations (1):
- VA Puget Sound Health Care System Seattle Division, Seattle, WA, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
Only completely deidentified/anonymized versions of datasets would be shared, provided that appropriate enterprise-level procedures permit this and are in place. Sharing would only take place under a written agreement prohibiting the recipient from identifying or re-identifying (or taking steps to identify or re-identify) any individual whose data are included in the dataset, including a properly submitted FOIA request. Electronic versions of final data sets will be maintained locally in a secure manner until enterprise-level resources become available for long-term storage.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: The investigators will endeavor to share IPD when requested by 6 months after the time of publication of the main study findings and publication of longer-term results of the study, provided that appropriate enterprise-level procedures permit this and are in place at the time of.
Access Criteria: The study team and PI will review each request for IPD, with involvement of local administrative officials as appropriate. Requests will be evaluated for criteria including data safety, the purpose of analyses warranting potential risks of transferring data, security of the transfer. An agreement will specify the duration of time for data to be held before being destroyed at the destination site.

REFERENCES:
- [Derived] Tanus AD, Nishio I, Williams R, Friedly J, Soares B, Anderson D, Bambara J, Dawson T, Hsu A, Kim PY, Krashin D, Del Piero L, Korpak A, Timmons A, Suri P. Combining procedural and behavioral treatments for chronic low back pain: A pilot feasibility randomized controlled trial. PM R. 2025 Apr;17(4):431-444. doi: 10.1002/pmrj.13323. Epub 2025 Feb 4. PMID 39902653

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment dates: 11/15/2018 to 03/17/2020 at the VA Puget Sound Health Care System
Pre-assignment Details: The post-enrollment, pre-randomization run-in period was designed to exclude subjects who no longer met study criteria by the day of randomization, and those who were unlikely to be able to complete the study processes such as the telephone assessments used for data collection and the use of technology (synchronizing activity trackers).
Groups:
- Pre-Randomization Run-In Period: The pre-randomization run-in period was designed to exclude subjects who no longer met study criteria by the day of randomization, and those who were unlikely to be able to complete the study processes such as the telephone assessments used for data collection and the use of technology (synchronizing activity trackers). Of those who began the run-in period (n=16), 3 were withdrawn during the run-in period and prior to randomization, leaving 13 who were randomized.
- Group A (Lumbar Medial Branch Nerve Radiofrequency Ablation [LRFA] + AcTIVE-CBT): Participants received both:
  1. Lumbar medial branch nerve radiofrequency ablation (LRFA): Radiofrequency ablation of the dorsal rami of the lumbar spinal nerves, using electrode placement parallel to the medial branches, 18G electrodes or larger, and 2 lesions per nerve.
     and
  2. Activity-Tracker Informed Video-enabled Cognitive Behavioral Therapy (AcTIVE-CBT): AcTIVE-CBT involves a standardized CBT protocol for pain, delivered via a video telehealth interface. AcTIVE-CBT also incorporates use of an activity tracker to provide objective feedback on activity levels, which can inform participants' and providers' impressions of goals and progress.
- Group B (Simulated Lumbar Radiofrequency Ablation [Simulated LRFA] + AcTIVE-CBT): Participants received both:
  1. Simulated radiofrequency ablation of the dorsal rami of the lumbar spinal nerves (simulated LRFA), with targeted steroid injections: Performed in an identical fashion to the experimental arm (LRFA), except for medial branch lesioning, which will not be done in simulated LRFA, and 2) the simulated LRFA control group will receive an injection of triamcinolone acetonide at each site where a radiofrequency lesion would normally be applied.
     and
  2. Activity-Tracker Informed Video-enabled Cognitive Behavioral Therapy (AcTIVE-CBT): AcTIVE-CBT involves a standardized CBT protocol for pain, delivered via a video telehealth interface. AcTIVE-CBT also incorporates use of an activity tracker to provide objective feedback on activity levels, which can inform participants' and providers' impressions of goals and progress.
- Group C (Lumbar Medial Branch Nerve Radiofrequency Ablation [LRFA] + TBSCE): Participants received both:
  1. Lumbar medial branch nerve radiofrequency ablation (LRFA): Radiofrequency ablation of the dorsal rami of the lumbar spinal nerves, using electrode placement parallel to the medial branches, 18G electrodes or larger, and 2 lesions per nerve.
     and
  2. Telephone-based self-directed CBT and education (TBSCE): TBSCE control is a focused program of CBT involving an initial 60-minute telephone education session by a psychologist; the provision of printed educational materials on chronic pain self-management, and a workbook for CBT self-management; and structured, written plans for weekly practice, reading and homework using the workbook.
- Group D (Simulated Lumbar Radiofrequency Ablation [Simulated LRFA] + TBSCE): Participants received both:
  1. Simulated radiofrequency ablation of the dorsal rami of the lumbar spinal nerves (simulated LRFA), with targeted steroid injections: Performed in an identical fashion to the experimental arm (LRFA), except for medial branch lesioning, which will not be done in simulated LRFA, and the simulated LRFA control group will receive an injection of triamcinolone acetonide at each site where a radiofrequency lesion would normally be applied.
     and
  2. Telephone-based self-directed CBT and education (TBSCE): TBSCE control is a focused program of CBT involving an initial 60-minute telephone education session by a psychologist; the provision of printed educational materials on chronic pain self-management, and a workbook for CBT self-management; and structured, written plans for weekly practice, reading and homework using the workbook.
Period: Pre-Randomization
Arm/Group | Pre-Randomization Run-In Period | Group A (Lumbar Medial Branch Nerve Radiofrequency Ablation [LRFA] + AcTIVE-CBT) | Group B (Simulated Lumbar Radiofrequency Ablation [Simulated LRFA] + AcTIVE-CBT) | Group C (Lumbar Medial Branch Nerve Radiofrequency Ablation [LRFA] + TBSCE) | Group D (Simulated Lumbar Radiofrequency Ablation [Simulated LRFA] + TBSCE)
Started | 16 | 0 (Although participant flow is presented for each cell of the 2 x 2 contingency table in this factorial pilot trial, the primary analysis as originally planned focused on the main effects of (1) LRFA vs. simulated LRFA and (2) AcTIVE-CBT vs. TBSCE, unless there were indications of strong interactions between the two types of treatment. There are no participants in this group until the randomization period (until after the pre-randomization run-in period has ended).) | 0 (Although participant flow is presented for each cell of the 2 x 2 contingency table in this factorial pilot trial, the primary analysis as originally planned focused on the main effects of (1) LRFA vs. simulated LRFA and (2) AcTIVE-CBT vs. TBSCE, unless there were indications of strong interactions between the two types of treatment. There are no participants in this group until the randomization period (until after the pre-randomization run-in period has ended).) | 0 (Although participant flow is presented for each cell of the 2 x 2 contingency table in this factorial pilot trial, the primary analysis as originally planned focused on the main effects of (1) LRFA vs. simulated LRFA and (2) AcTIVE-CBT vs. TBSCE, unless there were indications of strong interactions between the two types of treatment. There are no participants in this group until the randomization period (until after the pre-randomization run-in period has ended).) | 0 (Although participant flow is presented for each cell of the 2 x 2 contingency table in this factorial pilot trial, the primary analysis as originally planned focused on the main effects of (1) LRFA vs. simulated LRFA and (2) AcTIVE-CBT vs. TBSCE, unless there were indications of strong interactions between the two types of treatment. There are no participants in this group until the randomization period (until after the pre-randomization run-in period has ended).)
Completed | 13 | 0 | 0 | 0 | 0
Not Completed | 3 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0
Not completed — Failed eligibility criteria or run-in period criteria | 2 | 0 | 0 | 0 | 0
Period: Randomized
Arm/Group | Pre-Randomization Run-In Period | Group A (Lumbar Medial Branch Nerve Radiofrequency Ablation [LRFA] + AcTIVE-CBT) | Group B (Simulated Lumbar Radiofrequency Ablation [Simulated LRFA] + AcTIVE-CBT) | Group C (Lumbar Medial Branch Nerve Radiofrequency Ablation [LRFA] + TBSCE) | Group D (Simulated Lumbar Radiofrequency Ablation [Simulated LRFA] + TBSCE)
Started | 0 (There are no participants in this group during this period, because the pre-randomization run-in period has ended.) | 4 (Although participant flow is presented for each cell of the 2 x 2 contingency table in this factorial pilot trial, the primary analysis as originally planned focused on the main effects of (1) LRFA vs. simulated LRFA and (2) AcTIVE-CBT vs. TBSCE, unless there were indications of strong interactions between the two types of treatment.) | 3 (Although participant flow is presented for each cell of the 2 x 2 contingency table in this factorial pilot trial, the primary analysis as originally planned focused on the main effects of (1) LRFA vs. simulated LRFA and (2) AcTIVE-CBT vs. TBSCE, unless there were indications of strong interactions between the two types of treatment.) | 3 (Although participant flow is presented for each cell of the 2 x 2 contingency table in this factorial pilot trial, the primary analysis as originally planned focused on the main effects of (1) LRFA vs. simulated LRFA and (2) AcTIVE-CBT vs. TBSCE, unless there were indications of strong interactions between the two types of treatment.) | 3 (Although participant flow is presented for each cell of the 2 x 2 contingency table in this factorial pilot trial, the primary analysis as originally planned focused on the main effects of (1) LRFA vs. simulated LRFA and (2) AcTIVE-CBT vs. TBSCE, unless there were indications of strong interactions between the two types of treatment.)
Completed | 0 | 4 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: At randomization, participants are randomized to 1 the 4 treatment groups above; thus there are 0 participants in the "Pre-Randomization Run-In Period" group. Although baseline characteristics presented for each cell of the 2 x 2 contingency table in this factorial pilot trial, the primary analysis as originally planned focused on the main effects of (1) LRFA vs. simulated LRFA and (2) AcTIVE-CBT vs. TBSCE, unless there were indications of strong interactions between the two types of treatment.
Groups:
- Pre-Randomization Run-In Period: The pre-randomization run-in period was designed to exclude subjects who no longer met study criteria by the day of randomization, and those who were unlikely to be able to complete the study processes such as the telephone assessments used for data collection and the use of technology (synchronizing activity trackers). Of those who began the run-in period (n=16), 3 were withdrawn during the run-in period and prior to randomization, leaving 13 who were randomized. There are no participants in this group after randomization.
- Lumbar Medial Branch Nerve Radiofrequency Ablation (LRFA) + AcTIVE-CBT: Participants received both:
  1. Lumbar medial branch nerve radiofrequency ablation (LRFA): Radiofrequency ablation of the dorsal rami of the lumbar spinal nerves, using electrode placement parallel to the medial branches, 18G electrodes or larger, and 2 lesions per nerve.
     and
  2. Activity-Tracker Informed Video-enabled Cognitive Behavioral Therapy (AcTIVE-CBT): AcTIVE-CBT involves a standardized CBT protocol for pain, delivered via a video telehealth interface. AcTIVE-CBT also incorporates use of an activity tracker to provide objective feedback on activity levels, which can inform participants' and providers' impressions of goals and progress.
- Simulated Lumbar Radiofrequency Ablation (Simulated LRFA) + AcTIVE-CBT: Participants received both:
  1. Simulated radiofrequency ablation of the dorsal rami of the lumbar spinal nerves (simulated LRFA), with targeted steroid injections: Performed in an identical fashion to the experimental arm (LRFA), except for medial branch lesioning, which will not be done in simulated LRFA, and 2) the simulated LRFA control group will receive an injection of triamcinolone acetonide at each site where a radiofrequency lesion would normally be applied.
     and
  2. Activity-Tracker Informed Video-enabled Cognitive Behavioral Therapy (AcTIVE-CBT): AcTIVE-CBT involves a standardized CBT protocol for pain, delivered via a video telehealth interface. AcTIVE-CBT also incorporates use of an activity tracker to provide objective feedback on activity levels, which can inform participants' and providers' impressions of goals and progress.
- Lumbar Medial Branch Nerve Radiofrequency Ablation (LRFA) + TBSCE: Participants received both:
  1. Lumbar medial branch nerve radiofrequency ablation (LRFA): Radiofrequency ablation of the dorsal rami of the lumbar spinal nerves, using electrode placement parallel to the medial branches, 18G electrodes or larger, and 2 lesions per nerve.
     and
  2. Telephone-based self-directed CBT and education (TBSCE): TBSCE control is a focused program of CBT involving an initial 60-minute telephone education session by a psychologist; the provision of printed educational materials on chronic pain self-management, and a workbook for CBT self-management; and structured, written plans for weekly practice, reading and homework using the workbook.
- Simulated Lumbar Radiofrequency Ablation (Simulated LRFA) + TBSCE: Participants received both:
  1. Simulated radiofrequency ablation of the dorsal rami of the lumbar spinal nerves (simulated LRFA), with targeted steroid injections: Performed in an identical fashion to the experimental arm (LRFA), except for medial branch lesioning, which will not be done in simulated LRFA, and the simulated LRFA control group will receive an injection of triamcinolone acetonide at each site where a radiofrequency lesion would normally be applied.
     and
  2. Telephone-based self-directed CBT and education (TBSCE): TBSCE control is a focused program of CBT involving an initial 60-minute telephone education session by a psychologist; the provision of printed educational materials on chronic pain self-management, and a workbook for CBT self-management; and structured, written plans for weekly practice, reading and homework using the workbook.
- Total: Total of all reporting groups
Arm/Group | Pre-Randomization Run-In Period | Lumbar Medial Branch Nerve Radiofrequency Ablation (LRFA) + AcTIVE-CBT | Simulated Lumbar Radiofrequency Ablation (Simulated LRFA) + AcTIVE-CBT | Lumbar Medial Branch Nerve Radiofrequency Ablation (LRFA) + TBSCE | Simulated Lumbar Radiofrequency Ablation (Simulated LRFA) + TBSCE | Total
Number analyzed (Participants) | 0 | 4 | 3 | 3 | 3 | 13
Age, Continuous [Mean (Standard Deviation); unit: years] |  | 59.3 (14.6) | 57.7 (14.6) | 66.0 (14.1) | 49.3 (3.5) | 58.2 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female |  | 0 | 0 | 0 | 0 | 0
  Male |  | 4 | 3 | 3 | 3 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino |  | 2 | 1 | 0 | 0 | 3
  Not Hispanic or Latino |  | 2 | 2 | 3 | 3 | 10
  Unknown or Not Reported |  | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native |  | 0 | 0 | 0 | 0 | 0
  Asian |  | 0 | 2 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander |  | 0 | 0 | 0 | 0 | 0
  Black or African American |  | 0 | 0 | 0 | 0 | 0
  White |  | 3 | 1 | 2 | 3 | 9
  More than one race |  | 0 | 0 | 1 | 0 | 1
  Unknown or Not Reported |  | 1 | 0 | 0 | 0 | 1
Back-related functional limitations, RMDQ (pre-randomization) [Mean (Standard Deviation); unit: units on a scale] — The Roland-Morris Disability Questionnaire (RMDQ) is a validated, commonly used, and widely accepted measure of back-related functional limitations. Scores range from 0 to 24, with higher numbers reflecting greater functional limitations.
  units on a scale |  | 16.3 (3.6) | 10.0 (3.6) | 14.0 (1.0) | 16.0 (2.7) | 14.2 (3.7)

OUTCOME MEASURES:

1. Primary Outcome: Roland-Morris Disability Questionnaire
Description: The RMDQ is a validated, commonly used, and widely accepted 'legacy' measure of back-related functional limitations (range 0 to 24, with higher scores representing greater functional limitations).
Time Frame: 3 months
Population: Note that this outcome reporting does not include the "Pre-Randomization Run-In Period Arm/Group", because that group is not mutually exclusive from the 4 groups presented here (it includes the same participants, but prior to randomization).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group A (Lumbar Medial Branch Nerve Radiofrequency Ablation [LRFA] + AcTIVE-CBT) | Group B (Simulated Lumbar Radiofrequency Ablation [Simulated LRFA] + AcTIVE-CBT) | Group C (Lumbar Medial Branch Nerve Radiofrequency Ablation [LRFA] + TBSCE) | Group D (Simulated Lumbar Radiofrequency Ablation [Simulated LRFA] + TBSCE)
Number analyzed (Participants) | 4 | 3 | 3 | 3
units on a scale | 9.8 (4.1) | 5.3 (5.9) | 13.3 (3.1) | 16.7 (4.2)
Statistical Analysis 1: Comparison: Group A (Lumbar Medial Branch Nerve Radiofrequency Ablation [LRFA] + AcTIVE-CBT) vs Group B (Simulated Lumbar Radiofrequency Ablation [Simulated LRFA] + AcTIVE-CBT) vs Group C (Lumbar Medial Branch Nerve Radiofrequency Ablation [LRFA] + TBSCE) vs Group D (Simulated Lumbar Radiofrequency Ablation [Simulated LRFA] + TBSCE); Test type: Superiority; Mean Difference (Final Values) = -3.3, 95% CI 2-sided [-10.2 to 3.7], Standard Error of Mean 3.1 — Analysis of the MAIN EFFECT of LRFA (Group A + Group C) vs. simulated LRFA (Group B + Group D) on the outcome at 3 months, after adjustment for age and baseline value of the outcome. Negative scores indicate benefit with LRFA over simulated LRFA
Statistical Analysis 2: Comparison: Group A (Lumbar Medial Branch Nerve Radiofrequency Ablation [LRFA] + AcTIVE-CBT) vs Group B (Simulated Lumbar Radiofrequency Ablation [Simulated LRFA] + AcTIVE-CBT) vs Group C (Lumbar Medial Branch Nerve Radiofrequency Ablation [LRFA] + TBSCE) vs Group D (Simulated Lumbar Radiofrequency Ablation [Simulated LRFA] + TBSCE); Test type: Superiority; Mean Difference (Final Values) = -6.3, 95% CI 2-sided [-11.0 to -1.6], Standard Error of Mean 2.1 — Analysis of the MAIN EFFECT of AcTIVE-CBT (Group A + Group B) vs. TBSCE (Group C + Group D) on the outcome at 3 months, after adjustment for age and baseline value of the outcome. Negative scores indicate benefit with AcTIVE-CBT over TBSCE

2. Secondary Outcome: Activity Tracker-assessed Average Daily Step Counts (Change Scores)
Description: Change scores will be calculated as compared to average daily step count pre-randomization.
Time Frame: 3 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: average daily step count change score
Arm/Group | Group A (Lumbar Medial Branch Nerve Radiofrequency Ablation [LRFA] + AcTIVE-CBT) | Group B (Simulated Lumbar Radiofrequency Ablation [Simulated LRFA] + AcTIVE-CBT) | Group C (Lumbar Medial Branch Nerve Radiofrequency Ablation [LRFA] + TBSCE) | Group D (Simulated Lumbar Radiofrequency Ablation [Simulated LRFA] + TBSCE)
Number analyzed (Participants) | 4 | 3 | 3 | 3
average daily step count change score | -1445.8 (5984.0) | 5617.2 (5963.4) | 42.02 (448.3) | -842.4 (3105.5)
Statistical Analysis 1: Comparison: Group A (Lumbar Medial Branch Nerve Radiofrequency Ablation [LRFA] + AcTIVE-CBT) vs Group B (Simulated Lumbar Radiofrequency Ablation [Simulated LRFA] + AcTIVE-CBT) vs Group C (Lumbar Medial Branch Nerve Radiofrequency Ablation [LRFA] + TBSCE) vs Group D (Simulated Lumbar Radiofrequency Ablation [Simulated LRFA] + TBSCE); Test type: Superiority; Mean Difference (Final Values) = -6059.0, 95% CI 2-sided [-12467.0 to 349.1], Standard Error of Mean 2832.7 — This is an analysis of the MAIN EFFECT of LRFA (Group A + Group C) vs. simulated LRFA (Group B + Group D) on CHANGE in step counts, after adjustment for age and baseline step counts. Positive values show increased steps with LRFA over simulated LRFA
Statistical Analysis 2: Comparison: Group A (Lumbar Medial Branch Nerve Radiofrequency Ablation [LRFA] + AcTIVE-CBT) vs Group B (Simulated Lumbar Radiofrequency Ablation [Simulated LRFA] + AcTIVE-CBT) vs Group C (Lumbar Medial Branch Nerve Radiofrequency Ablation [LRFA] + TBSCE) vs Group D (Simulated Lumbar Radiofrequency Ablation [Simulated LRFA] + TBSCE); Test type: Superiority; Mean Difference (Final Values) = 2081.9, 95% CI 2-sided [-4666.6 to 8830.4], Standard Error of Mean 2983.2 — This is an analysis of the MAIN EFFECT of AcTIVE-CBT (Group A + Group B) vs. TBSCE (Group C + Group D) on CHANGE in step counts, after adjustment for age and baseline step counts.Positive values show increased steps with AcTIVE-CBT over TBSCE

3. Secondary Outcome: Low Back Pain Intensity (0-10 Numerical Pain Rating Scale)
Description: Higher numerical pain ratings reflect greater pain intensity.
Time Frame: 3 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group A (Lumbar Medial Branch Nerve Radiofrequency Ablation [LRFA] + AcTIVE-CBT) | Group B (Simulated Lumbar Radiofrequency Ablation [Simulated LRFA] + AcTIVE-CBT) | Group C (Lumbar Medial Branch Nerve Radiofrequency Ablation [LRFA] + TBSCE) | Group D (Simulated Lumbar Radiofrequency Ablation [Simulated LRFA] + TBSCE)
Number analyzed (Participants) | 4 | 3 | 3 | 3
units on a scale | 4.8 (4.5) | 4.7 (1.2) | 4.7 (3.5) | 5.3 (1.5)
Statistical Analysis 1: Comparison: Group A (Lumbar Medial Branch Nerve Radiofrequency Ablation [LRFA] + AcTIVE-CBT) vs Group B (Simulated Lumbar Radiofrequency Ablation [Simulated LRFA] + AcTIVE-CBT) vs Group C (Lumbar Medial Branch Nerve Radiofrequency Ablation [LRFA] + TBSCE) vs Group D (Simulated Lumbar Radiofrequency Ablation [Simulated LRFA] + TBSCE); Test type: Superiority; Mean Difference (Final Values) = -1.0, 95% CI 2-sided [-5.2 to 3.1], Standard Error of Mean 1.8 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Group A (Lumbar Medial Branch Nerve Radiofrequency Ablation [LRFA] + AcTIVE-CBT) vs Group B (Simulated Lumbar Radiofrequency Ablation [Simulated LRFA] + AcTIVE-CBT) vs Group C (Lumbar Medial Branch Nerve Radiofrequency Ablation [LRFA] + TBSCE) vs Group D (Simulated Lumbar Radiofrequency Ablation [Simulated LRFA] + TBSCE); Test type: Superiority; Mean Difference (Final Values) = -0.3, 95% CI 2-sided [-4.2 to 3.6], Standard Error of Mean 1.7 — [estimate comment as in outcome 1, analysis 2]

4. Secondary Outcome: PROMIS Global Health Short Form 10
Description: Global quality of life measure. There are two subscales, the physical component summary score and the mental component summary score. Each range from 4-20, with higher scores reflecting greater quality of life
Time Frame: 3 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group A (Lumbar Medial Branch Nerve Radiofrequency Ablation [LRFA] + AcTIVE-CBT) | Group B (Simulated Lumbar Radiofrequency Ablation [Simulated LRFA] + AcTIVE-CBT) | Group C (Lumbar Medial Branch Nerve Radiofrequency Ablation [LRFA] + TBSCE) | Group D (Simulated Lumbar Radiofrequency Ablation [Simulated LRFA] + TBSCE)
Number analyzed (Participants) | 4 | 3 | 3 | 3
units on a scale
  PROMIS physical health | 40.5 (5.2) | 44.3 (5.8) | 37.4 (9.3) | 38.2 (3.8)
  PROMIS mental health | 47.8 (5.4) | 50.9 (5.1) | 55.3 (4.2) | 38.6 (7.3)
Statistical Analysis 1: Comparison: Group A (Lumbar Medial Branch Nerve Radiofrequency Ablation [LRFA] + AcTIVE-CBT) vs Group B (Simulated Lumbar Radiofrequency Ablation [Simulated LRFA] + AcTIVE-CBT) vs Group C (Lumbar Medial Branch Nerve Radiofrequency Ablation [LRFA] + TBSCE) vs Group D (Simulated Lumbar Radiofrequency Ablation [Simulated LRFA] + TBSCE); PROMIS physical health scores; Test type: Superiority; Mean Difference (Final Values) = 1.0, 95% CI 2-sided [-8.1 to 10.1], Standard Error of Mean 4.0 — Analysis of the MAIN EFFECT of LRFA (Group A + Group C) vs. simulated LRFA (Group B + Group D) on the outcome at 3 months after adjustment for age and baseline value of the outcome. Positive scores indicate better health with LRFA vs. simulated LRFA
Statistical Analysis 2: Comparison: Group A (Lumbar Medial Branch Nerve Radiofrequency Ablation [LRFA] + AcTIVE-CBT) vs Group B (Simulated Lumbar Radiofrequency Ablation [Simulated LRFA] + AcTIVE-CBT) vs Group C (Lumbar Medial Branch Nerve Radiofrequency Ablation [LRFA] + TBSCE) vs Group D (Simulated Lumbar Radiofrequency Ablation [Simulated LRFA] + TBSCE); PROMIS physical health scores; Test type: Superiority; Mean Difference (Final Values) = 6.2, 95% CI 2-sided [-0.4 to 12.9], Standard Error of Mean 2.9 — Analysis of the MAIN EFFECT of AcTIVE-CBT (Group A + Group B) vs. TBSCE (Group C + Group D) on the outcome at 3 months after adjustment for age and baseline value of the outcome. Positive scores indicate better health with AcTIVE-CBT vs. TBSCE
Statistical Analysis 3: Comparison: Group A (Lumbar Medial Branch Nerve Radiofrequency Ablation [LRFA] + AcTIVE-CBT) vs Group B (Simulated Lumbar Radiofrequency Ablation [Simulated LRFA] + AcTIVE-CBT) vs Group C (Lumbar Medial Branch Nerve Radiofrequency Ablation [LRFA] + TBSCE) vs Group D (Simulated Lumbar Radiofrequency Ablation [Simulated LRFA] + TBSCE); PROMIS mental health scores; Test type: Superiority; Mean Difference (Final Values) = 3.7, 95% CI 2-sided [-5.4 to 12.7], Standard Error of Mean 4.0 — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 4: Comparison: Group A (Lumbar Medial Branch Nerve Radiofrequency Ablation [LRFA] + AcTIVE-CBT) vs Group B (Simulated Lumbar Radiofrequency Ablation [Simulated LRFA] + AcTIVE-CBT) vs Group C (Lumbar Medial Branch Nerve Radiofrequency Ablation [LRFA] + TBSCE) vs Group D (Simulated Lumbar Radiofrequency Ablation [Simulated LRFA] + TBSCE); PROMIS mental health scores; Test type: Superiority; Mean Difference (Final Values) = 1.8, 95% CI 2-sided [-7.0 to 10.6], Standard Error of Mean 3.9 — [estimate comment as in outcome 4, analysis 2]

5. Secondary Outcome: Average Morphine Equivalent Daily Dose
Description: Self-reported average morphine equivalent daily dose over the past 3 days.
Time Frame: 3 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: average morphine milligram equivalents
Arm/Group | Group A (Lumbar Medial Branch Nerve Radiofrequency Ablation [LRFA] + AcTIVE-CBT) | Group B (Simulated Lumbar Radiofrequency Ablation [Simulated LRFA] + AcTIVE-CBT) | Group C (Lumbar Medial Branch Nerve Radiofrequency Ablation [LRFA] + TBSCE) | Group D (Simulated Lumbar Radiofrequency Ablation [Simulated LRFA] + TBSCE)
Number analyzed (Participants) | 4 | 3 | 3 | 3
average morphine milligram equivalents | 0 (0) | 0 (0) | 0 (0) | 6.7 (5.8)
Statistical Analysis 1: Comparison: Group A (Lumbar Medial Branch Nerve Radiofrequency Ablation [LRFA] + AcTIVE-CBT) vs Group B (Simulated Lumbar Radiofrequency Ablation [Simulated LRFA] + AcTIVE-CBT) vs Group C (Lumbar Medial Branch Nerve Radiofrequency Ablation [LRFA] + TBSCE) vs Group D (Simulated Lumbar Radiofrequency Ablation [Simulated LRFA] + TBSCE); Test type: Superiority; Mean Difference (Final Values) = -2.9, 95% CI 2-sided [-7.7 to 1.9], Standard Error of Mean 2.1 — Analysis of the MAIN EFFECT of LRFA (Group A + Group C) vs. simulated LRFA (Group B + Group D) on the outcome at 3 months, after adjustment for age and baseline value of the outcome. Negative scores indicate lower doses with LRFA over simulated LRFA
Statistical Analysis 2: Comparison: Group A (Lumbar Medial Branch Nerve Radiofrequency Ablation [LRFA] + AcTIVE-CBT) vs Group B (Simulated Lumbar Radiofrequency Ablation [Simulated LRFA] + AcTIVE-CBT) vs Group C (Lumbar Medial Branch Nerve Radiofrequency Ablation [LRFA] + TBSCE) vs Group D (Simulated Lumbar Radiofrequency Ablation [Simulated LRFA] + TBSCE); Test type: Superiority; Mean Difference (Final Values) = -3.3, 95% CI 2-sided [-7.5 to 1.0], Standard Error of Mean 1.9 — Analysis of the MAIN EFFECT of AcTIVE-CBT (Group A + Group B) vs. TBSCE (Group C + Group D) on the outcome at 3 months, after adjustment for age and baseline value of the outcome. Negative scores indicate lower doses with AcTIVE-CBT over TBSCE

6. Secondary Outcome: Global Perceived Effect (How Back Pain Has Changed Since Baseline)
Description: 7-point Likert scale where 3 represents 'complete recovery', 0 represents 'not changed', and -3 represents 'become worse than ever'
Time Frame: 3 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group A (Lumbar Medial Branch Nerve Radiofrequency Ablation [LRFA] + AcTIVE-CBT) | Group B (Simulated Lumbar Radiofrequency Ablation [Simulated LRFA] + AcTIVE-CBT) | Group C (Lumbar Medial Branch Nerve Radiofrequency Ablation [LRFA] + TBSCE) | Group D (Simulated Lumbar Radiofrequency Ablation [Simulated LRFA] + TBSCE)
Number analyzed (Participants) | 4 | 3 | 3 | 3
units on a scale | 0.3 (1.7) | 0.7 (0.6) | 0.7 (1.2) | 0 (0)
Statistical Analysis 1: Comparison: Group A (Lumbar Medial Branch Nerve Radiofrequency Ablation [LRFA] + AcTIVE-CBT) vs Group B (Simulated Lumbar Radiofrequency Ablation [Simulated LRFA] + AcTIVE-CBT) vs Group C (Lumbar Medial Branch Nerve Radiofrequency Ablation [LRFA] + TBSCE) vs Group D (Simulated Lumbar Radiofrequency Ablation [Simulated LRFA] + TBSCE); Test type: Superiority; Mean Difference (Final Values) = 0.2, 95% CI 2-sided [-1.4 to 1.7], Standard Error of Mean 0.7 — Analysis of the MAIN EFFECT of LRFA (Group A + Group C) vs. simulated LRFA (Group B + Group D) on the outcome at 3 months, after adjustment for age. Positive scores indicate perceived benefit with LRFA over simulated LRFA
Statistical Analysis 2: Comparison: Group A (Lumbar Medial Branch Nerve Radiofrequency Ablation [LRFA] + AcTIVE-CBT) vs Group B (Simulated Lumbar Radiofrequency Ablation [Simulated LRFA] + AcTIVE-CBT) vs Group C (Lumbar Medial Branch Nerve Radiofrequency Ablation [LRFA] + TBSCE) vs Group D (Simulated Lumbar Radiofrequency Ablation [Simulated LRFA] + TBSCE); Test type: Superiority; Mean Difference (Final Values) = 0.1, 95% CI 2-sided [-1.3 to 1.5], Standard Error of Mean 0.6 — Analysis of the MAIN EFFECT of AcTIVE-CBT (Group A + Group B) vs. TBSCE (Group C + Group D) on the outcome at 3 months, after adjustment for age and baseline value of the outcome. Positive scores indicate perceived benefit with AcTIVE-CBT over TBSCE

7. Secondary Outcome: Expected Low Back Pain Intensity (0-10 Numerical Pain Rating Scale) if Not Using Pain Medications
Description: Higher numerical pain ratings reflect greater pain intensity.
Time Frame: 3 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group A (Lumbar Medial Branch Nerve Radiofrequency Ablation [LRFA] + AcTIVE-CBT) | Group B (Simulated Lumbar Radiofrequency Ablation [Simulated LRFA] + AcTIVE-CBT) | Group C (Lumbar Medial Branch Nerve Radiofrequency Ablation [LRFA] + TBSCE) | Group D (Simulated Lumbar Radiofrequency Ablation [Simulated LRFA] + TBSCE)
Number analyzed (Participants) | 4 | 3 | 3 | 3
units on a scale | 5.0 (4.2) | 5.0 (1.7) | 5.7 (4.0) | 7.0 (1.7)
Statistical Analysis 1: Comparison: Group A (Lumbar Medial Branch Nerve Radiofrequency Ablation [LRFA] + AcTIVE-CBT) vs Group B (Simulated Lumbar Radiofrequency Ablation [Simulated LRFA] + AcTIVE-CBT) vs Group C (Lumbar Medial Branch Nerve Radiofrequency Ablation [LRFA] + TBSCE) vs Group D (Simulated Lumbar Radiofrequency Ablation [Simulated LRFA] + TBSCE); Test type: Superiority; Mean Difference (Final Values) = -0.9, 95% CI 2-sided [-5.5 to 3.7], Standard Error of Mean 2.0 — Analysis of the MAIN EFFECT of LRFA (Group A + Group C) vs. simulated LRFA (Group B + Group D) on the outcome at 3 months after adjustment for age and baseline value of the outcome. Negative scores indicate less pain with LRFA over simulated LRFA
Statistical Analysis 2: Comparison: Group A (Lumbar Medial Branch Nerve Radiofrequency Ablation [LRFA] + AcTIVE-CBT) vs Group B (Simulated Lumbar Radiofrequency Ablation [Simulated LRFA] + AcTIVE-CBT) vs Group C (Lumbar Medial Branch Nerve Radiofrequency Ablation [LRFA] + TBSCE) vs Group D (Simulated Lumbar Radiofrequency Ablation [Simulated LRFA] + TBSCE); Test type: Superiority; Mean Difference (Final Values) = -1.4, 95% CI 2-sided [-5.4 to 2.6], Standard Error of Mean 1.8 — Analysis of the MAIN EFFECT of AcTIVE-CBT (Group A + Group B) vs. TBSCE (Group C + Group D) on the outcome at 3 months after adjustment for age and baseline value of the outcome. Negative scores indicate less pain with AcTIVE-CBT vs. TBSCE

8. Secondary Outcome: Participant-reported Satisfaction
Description: 5-point Likert scale where 2 represents 'completely satisfied', 0 represents 'neutral', and -2 represents 'completely dissatisfied'
Time Frame: 3 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group A (Lumbar Medial Branch Nerve Radiofrequency Ablation [LRFA] + AcTIVE-CBT) | Group B (Simulated Lumbar Radiofrequency Ablation [Simulated LRFA] + AcTIVE-CBT) | Group C (Lumbar Medial Branch Nerve Radiofrequency Ablation [LRFA] + TBSCE) | Group D (Simulated Lumbar Radiofrequency Ablation [Simulated LRFA] + TBSCE)
Number analyzed (Participants) | 4 | 3 | 3 | 3
units on a scale | 1.0 (1.4) | 0.3 (0.6) | 0.3 (1.5) | -1.3 (0.6)
Statistical Analysis 1: Comparison: Group A (Lumbar Medial Branch Nerve Radiofrequency Ablation [LRFA] + AcTIVE-CBT) vs Group B (Simulated Lumbar Radiofrequency Ablation [Simulated LRFA] + AcTIVE-CBT) vs Group C (Lumbar Medial Branch Nerve Radiofrequency Ablation [LRFA] + TBSCE) vs Group D (Simulated Lumbar Radiofrequency Ablation [Simulated LRFA] + TBSCE); Test type: Superiority; Mean Difference (Final Values) = 1.3, 95% CI 2-sided [-0.5 to 3.0], Standard Error of Mean 0.8 — Analysis of the MAIN EFFECT of LRFA (Group A + Group C) vs. simulated LRFA (Group B + Group D) on the outcome at 3 months, after adjustment for age. Positive scores indicate more satisfaction with LRFA over simulated LRFA
Statistical Analysis 2: Comparison: Group A (Lumbar Medial Branch Nerve Radiofrequency Ablation [LRFA] + AcTIVE-CBT) vs Group B (Simulated Lumbar Radiofrequency Ablation [Simulated LRFA] + AcTIVE-CBT) vs Group C (Lumbar Medial Branch Nerve Radiofrequency Ablation [LRFA] + TBSCE) vs Group D (Simulated Lumbar Radiofrequency Ablation [Simulated LRFA] + TBSCE); Test type: Superiority; Mean Difference (Final Values) = 1.2, 95% CI 2-sided [-0.4 to 2.8], Standard Error of Mean 0.7 — Analysis of the MAIN EFFECT of AcTIVE-CBT (Group A + Group B) vs. TBSCE (Group C + Group D) on the outcome at 3 months, after adjustment for age. Positive scores indicate more satisfaction with AcTIVE-CBT over TBSCE

9. Secondary Outcome: BRFSS Self-reported Physical Activity Per Week
Description: Self-reported activity equivalent minutes per week
Time Frame: 3 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: activity minutes per week
Arm/Group | Group A (Lumbar Medial Branch Nerve Radiofrequency Ablation [LRFA] + AcTIVE-CBT) | Group B (Simulated Lumbar Radiofrequency Ablation [Simulated LRFA] + AcTIVE-CBT) | Group C (Lumbar Medial Branch Nerve Radiofrequency Ablation [LRFA] + TBSCE) | Group D (Simulated Lumbar Radiofrequency Ablation [Simulated LRFA] + TBSCE)
Number analyzed (Participants) | 4 | 3 | 3 | 3
activity minutes per week | 487.5 (306.2) | 1650.0 (297.0) | 201.7 (97.8) | 398.3 (530.1)
Statistical Analysis 1: Comparison: Group A (Lumbar Medial Branch Nerve Radiofrequency Ablation [LRFA] + AcTIVE-CBT) vs Group B (Simulated Lumbar Radiofrequency Ablation [Simulated LRFA] + AcTIVE-CBT) vs Group C (Lumbar Medial Branch Nerve Radiofrequency Ablation [LRFA] + TBSCE) vs Group D (Simulated Lumbar Radiofrequency Ablation [Simulated LRFA] + TBSCE); Test type: Superiority; Mean Difference (Final Values) = -637.0, 95% CI 2-sided [-1636.2 to 362.1], Standard Error of Mean 433.3 — Analysis of the MAIN EFFECT of LRFA (Group A + Group C) vs. simulated LRFA (Group B + Group D) on the outcome at 3 months adjusting for age and baseline value of the outcome. Positive scores indicate greater activity with LRFA over simulated LRFA
Statistical Analysis 2: Comparison: Group A (Lumbar Medial Branch Nerve Radiofrequency Ablation [LRFA] + AcTIVE-CBT) vs Group B (Simulated Lumbar Radiofrequency Ablation [Simulated LRFA] + AcTIVE-CBT) vs Group C (Lumbar Medial Branch Nerve Radiofrequency Ablation [LRFA] + TBSCE) vs Group D (Simulated Lumbar Radiofrequency Ablation [Simulated LRFA] + TBSCE); Test type: Superiority; Mean Difference (Final Values) = 572.2, 95% CI 2-sided [-199.3 to 1343.6], Standard Error of Mean 334.5 — Analysis of the MAIN EFFECT of AcTIVE-CBT (Group A + Group B) vs. TBSCE (Group C + Group D) on the outcome at 3 months adjusting for age and baseline value of the outcome. Positive scores indicate more satisfaction with AcTIVE-CBT over TBSCE

ADVERSE EVENTS:
Time Frame: 3 months
Description: Note that AE reporting includes the "Pre-Randomization Run-In Period Arm/Group", although that group is not mutually exclusive from the 4 groups presented here (it includes the same participants, but prior to randomization). We corresponded with the PRS Results Team who recommend this approach on 8/9/2021.
Groups:
- Pre-Randomizaton Run-In Period: The pre-randomization run-in period was designed to exclude subjects who no longer met study criteria by the day of randomization, and those who were unlikely to be able to complete the study processes such as the telephone assessments used for data collection and the use of technology (synchronizing activity trackers). Of those who began the run-in period (n=16), 3 were withdrawn during the run-in period and prior to randomization, leaving 13 who were randomized. There are no participants in this group after randomization.
Arm/Group | Pre-Randomizaton Run-In Period | Lumbar Medial Branch Nerve Radiofrequency Ablation (LRFA) + AcTIVE-CBT | Simulated Lumbar Radiofrequency Ablation (Simulated LRFA) + AcTIVE-CBT | Lumbar Medial Branch Nerve Radiofrequency Ablation (LRFA) + TBSCE | Simulated Lumbar Radiofrequency Ablation (Simulated LRFA) + TBSCE
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/4 | 0/3 | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/4 | 0/3 | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 5/16 | 3/4 | 1/3 | 3/3 | 0/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pre-Randomizaton Run-In Period (N=16) | Lumbar Medial Branch Nerve Radiofrequency Ablation (LRFA) + AcTIVE-CBT (N=4) | Simulated Lumbar Radiofrequency Ablation (Simulated LRFA) + AcTIVE-CBT (N=3) | Lumbar Medial Branch Nerve Radiofrequency Ablation (LRFA) + TBSCE (N=3) | Simulated Lumbar Radiofrequency Ablation (Simulated LRFA) + TBSCE (N=3)
Surgery (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ED/Urgent Care (Surgical and medical procedures) | 5 (5) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Hospitalization (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ICU (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Allergic Reaction (Immune system disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Other Complications (General disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-12): https://cdn.clinicaltrials.gov/large-docs/87/NCT03520387/Prot_SAP_000.pdf